CLINICAL TRIAL: NCT01872767
Title: Spectrum, Profile and Outcome of Infections in Patients With Cirrhosis and/ or Acute on Chronic Liver Failure Admitted in Liver Specialty ICU (Intensive Care Unit)- An Observational Study
Brief Title: Spectrum, Profile and Outcome of Infections in Patients With Cirrhosis and/ or Acute on Chronic Liver Failure
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-ACLF-0003
Record Dates: First submitted 2013-04-27; First posted 2013-06-07 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2014-11

CONDITIONS: Cirrhosis; Acute Liver Failure; Chronic Liver Failure
Keywords: Acute on Chronic Liver Failure (ACLF),Cirrhosis,; Institute of Liver & Biliary Sciences (ILBS)
MeSH Terms: conditions — Fibrosis; Liver Failure, Acute; End Stage Liver Disease; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cirrhotics/ Acute on chronic liver failure admitted to ICU

SUMMARY:
After successful screening diagnosis of cirrhosis and/or acute or chronic liver failure will be made. These patients will undergo detail clinical, biochemical and microbiological examination at baseline. Clinical examination and Biochemical evaluation will be done daily and signs of infection will be noted. Patients will undergo microbiological screening for infection every 48 hours. Patients suspected or diagnosed to be suffering from infections will be treated as per ILBS (Institute of Liver and Biliary Sciences) antibiotic policy. Site and etiology (bacterial and/or fungal) of infections will be noted in all patients at admission in liver specialty ICU (Intensive Care Unit) and during the ICU (Intensive Care Unit) stay. All the patients will be followed until discharge or death in ICU (Intensive Care Unit).

ELIGIBILITY:
Inclusion Criteria:

* A clinical, radiological or histological diagnosis of cirrhosis and/or ACLF (Acute on Chronic Liver Failure).
* Age > 18years

Exclusion Criteria:

* Previous liver transplantation.
* Patients who died within 8 hours of ICU (Intensive Care Unit) admission.
* Acute liver failure
* Lack of consent
* Patient on steroids/ or any other immunosuppressive medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary Care Center.
Sampling Method: Probability Sample
Enrollment: 522 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Mortality within 1 month during ICU (Intensive Care Unit) stay. | 30 days

SECONDARY OUTCOMES:
Number of days stayed in ICU (Intensive Care Unit). | 30 days
Risk factors determination in development of multidrug resistance bacteria.Risk factors are defined as Nosocomial infection,Recent Hospitalization, recent antibiotic usage, SBP (spontaneous bacterial peritonitis)prophylaxis, diabetes etc | 30 days
Proportion of patients with organ failure. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Amrish Sahney, MD, Principal Investigator — Institute of Liver & Biliary Sciences.
Locations (1):
- Institute of Liver & Biliary Sciences., New Delhi, National Capital Territory of Delhi, India